CLINICAL TRIAL: NCT04821479
Title: Safety and Clinical Effects of Repeated Intrathecal Injections of Autologous Mesenchymal Stem Cells in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Repeated Mesenchymal Stem Cell Injections in ALS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0208-16-HMO
Record Dates: First submitted 2020-10-19; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2020-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Mesenchymal stem cells; ALSFRSr
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — SLC25A33 protein, human

STUDY DESIGN:
Intervention Model Description: Single center open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repeated MSCs treatment in ALS patients (Experimental): Four intrathecal (IT) administrations of autologous MSC cells administered every 3 months in ALS patients. the IT treatment will be administered through a regular lumbar puncture at a dose of 1x10^6 MSCs per kg body weight in 3 ml saline.
  Interventions: Biological: Mesenchymal stem cells (MSC)

INTERVENTIONS:
Biological: Mesenchymal stem cells (MSC) — Intrathecal injections of autologous bone marrow derived mesenchymal stem cells
  Other Names: stem cells; Stromal cells

SUMMARY:
An open-label, single-center clinical trial to evaluate the safety and efficacy of repeated intrathecal administrations of autologous bone marrow derived mesenchyme stem cells in ALS patients. The study includes 20 subjects (age: 20-70) with definite diagnosis of ALS and ALS-FRS-R score of at least 20 and disease-duration of less than 3 years. The treatment protocol includes four intrathecal injections of MSC, at intervals of 3 months between the injections.

The primary endpoints are safety and tolerability. Several efficacy measures are assessed as secondary endpoints.

DETAILED DESCRIPTION:
An open-label, single-center clinical trial to evaluate the safety and efficacy of repeated intrathecal administrations of autologous bone marrow derived mesenchyme stem cells in ALS patients. The study includes 20 subjects (age: 20-70) with definite diagnosis of ALS and ALS-FRS-R score of at least 20 and disease-duration of less than 3 years. The treatment protocol includes four intrathecal injections of MSC, at intervals of 3 months between the injections. The primary endpoints are safety and tolerability. Several efficacy measures are assessed as secondary endpoints.

Applications from patients are received in our centre. An independent selective committee set by hospital's administration examines anonymously, according to the predefined inclusion and exclusion criteria. After inclusion and screening visit, patients are followed up for a "run-in" period of 6 months before the first visit (visit 1), to evaluate the progression rate of their disease. and for six months following the last transplantation.

One month after inclusion, patients undergo bone Marrow Aspiration (BMA) procedure and MSC cells are produced from the bone marrow aspirate. On the treatment visit, the patients are transplanted with an intrathecal (IT) injection of MSC (1 million cells per kg of body weight) and thereafter with additional injections every 3-6 months. After the MSC transplantation patients are examined on a bimonthly basis and evaluated for ALSFRSr scoring and forced vital capacity of the lungs (FVC) for a total follow up period of 3 months post last MSC-injection.

To establish the progression rate of the disease the monthly changes in the functional ALS score: ALSFRSr will be calculated during the 6 months-"run in period" and for the whole duration of the study, ending at 3 months following the last injection of MSC stem cells. The progression rate (as evidenced by the monthly changes in ALSFRSr and FVC) during the study (calculated at last visit time point, 3 months after the last MSC-injection) will be compared to the progression rate during the "run-in" period.

The follow up visits include observation for side effects, full neurological evaluation and muscle chart, ALS score and forced vital capacity (FVC) test. The safety is assessed following treatment with MSC, using measurements of the following variables: physical examination, vital signs (HR, BP, RR, body temperature), and clinical laboratory parameters: WBC with differential and platelet count, hemoglobin (Hb), hematocrit (Ht), blood chemistry for electrolytes, creatinine and liver enzymes.

All selected patients undergo bone marrow aspiration under light general anaesthesia and an inoculum of crude bone marrow cells (150 ml) is obtained and two thirds of it kept frozen. One third is cultured under GCP conditions at the human cell cultures clean room facility of Hadassah HMO. The MSCs are obtained from the bone marrow of each patient and prepared using our previously described protocol with slight modification.

One month later the patient is hospitalized and a lumbar puncture performed under standard conditions and local anaesthesia at the L4-5 lumbar level and 3 ml of CSF are removed and the cultured purified MSCs (1x106/kg of body weight) resuspended in 3 ml of normal saline are injected in the CSF, using a 20-gauge needle and 3-way cannula.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18 to 70 years old, at the Screening Visit.
2. Sporadic or familial ALS diagnosed patients fulfilling the El Escorial clinical criteria for definite.
3. Capable of providing informed consent and willing and able to follow study procedures, including willingness to undergo multiple/repeated lumbar punctures.
4. ALSFRS-R ≥15 at the Screening Visit.

Exclusion Criteria:

1. Patients with severe cognitive decline or inability to understand and sign the informed consent.
2. Participation in another clinical trial within 1 year prior to start of the study
3. Patients with active infections.
4. Positive test for Hepatitis B, Hepatitis C, and/or HIV per laboratory evaluations at the screening visit.
5. Any history of solid malignancy including any malignancy affecting the central nervous system within 5 years of the Screening Visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of multiple intrathecal MSC administration. Incidence of adverse events following multiple intrathecal MSC injections during 2 years follow-up period | Up to 18 months: starting from inclusion until 3 months after the last MSC-injection
  To evaluate the safety of 4 successive intrathecal administrations of autologous MSC cells administered every three months in ALS patient.
  Patients will be follow-up every 3 months for change in their neurological status and the incidence of adverse events. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Effect of repeated intrathecal MSC injections on the progression rate (monthly changes) of ALSFRSr | Up to 18 months: starting from inclusion until 3 months after the last MSC-injection.
  Degree of change in the rate of progression (calculation of monthly change in ALSFRSr score: 0-48, higher scores are better) between the run-in period to 3 months post last MSC-injection

SECONDARY OUTCOMES:
Effect of repeated intrathecal MSC injections on the progression rate (monthly changes) of respiratory forced vital capacity FVC | Up to 18 months: starting from inclusion until 3 months after the last MSC-injection.
  Degree of change in the rate of progression (calculation of monthly change in FVC score: 0-100%, higher numbers are better) between the run-in period to 3 months post last MSC-injection

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karussis, Professor, Principal Investigator — Hadassah HMO

REFERENCES:
- [Derived] Petrou P, Kassis I, Yaghmour NE, Ginzberg A, Karussis D. A phase II clinical trial with repeated intrathecal injections of autologous mesenchymal stem cells in patients with amyotrophic lateral sclerosis. Front Biosci (Landmark Ed). 2021 Oct 30;26(10):693-706. doi: 10.52586/4980. PMID 34719198